CLINICAL TRIAL: NCT05233527
Title: Observational, Retrospective, Monocentric Clinical Study on the Safety of Novosyn® Quick in Women With a Spontaneous Vaginal Delivery Who Required an Indicated Episiotomy
Brief Title: Novosyn® Quick in Patients Undergoing Episiotomy Closure
Acronym: RETRO-EPINOQ
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2111
Record Dates: First submitted 2022-01-26; First posted 2022-02-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Episiotomy Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Episiotomy Closure — indicated episiotomy with Novosyn® Quick after spontaneous vaginal delivery

SUMMARY:
Retrospective, monocentric clinical study on the clinical performance of Novosyn® Quick in patients undergoing episiotomy closure.

DETAILED DESCRIPTION:
The study design is a retrospective, consecutive series of women with a spontaneous vaginal delivery who required an indicated episiotomy with Novosyn® Quick between the period January 2020 - December 2020 at Hospital General de Catalunya.

All women treated with Novosyn® Quick between January 2020 - December 2020 at the Hospital General de Catalunya will be analyzed. The investigator team will access medical records for the cohort of patients identified.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent an indicated episiotomy between January 2020 - December 2020 at the Hospital General de Catalunya (Sant Cugat del Vallès, Spain) and received Novosyn® Quick

Exclusion Criteria:

* No exclusion criteria have been set

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with a spontaneous vaginal delivery who required an indicated episiotomy with Novosyn® Quick between the period January 2020 - December 2020 at Hospital General de Catalunya.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Wound dehiscence rate | up to 1 month postpartum
  A dehiscence of the wound which needs surgical treatment with re-closure.

SECONDARY OUTCOMES:
Rate of Re-suturing | up to 1 month postpartum
  Number of patients requiring a re-suturing due to wound dehiscence
Rate of Suture removal due to wound problems | up to 1 month postpartum
  Number of patients requiring suture removal due to wound problems (infection, gaping wound, residual material requiring removal)
Surgical Site Infection rate | up to 1 month postpartum
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections (A1) involving the skin only. Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material (A2).
Bleeding | up to 1 month postpartum
  Incidence of Bleeding after Episiotomy closure
Hematoma | up to 1 month postpartum
  Incidence of Hematoma after Episiotomy closure
Abscess formation | up to 1 month postpartum
  Incidence of Abscess formation after Episiotomy closure
Rectovaginal fistula | up to 1 month postpartum
  Incidence of Rectovaginal fistula after Episiotomy closure
Short-term perineal pain (VAS) | after 48 hours postpartum
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".
Long-term perineal pain (VAS) | up to 1 month postpartum
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".
Short-term Pain in daily living (VAS) | 24-48 hours postpartum
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".in repose, during walking, during sitting, when urinating, and when defecating
Long-term Pain in daily living (VAS) | up to 1 month postpartum
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".in repose, during walking, during sitting, when urinating, and when defecating

CONTACTS AND LOCATIONS:
Locations (1):
- IDC Hospital General de Catalunya, Sant Cugat del Vallès, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No